CLINICAL TRIAL: NCT06307379
Title: Patient Reported Outcome and Experience Measures for Bronchoscopic Procedures
Acronym: BRONCHOPROEM
Status: Recruiting | Type: Observational
Sponsor: Vitaz (Other)
Responsible Party: Sponsor
Other Study IDs: EC 23022
Record Dates: First submitted 2023-10-09; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Bronchial Diseases
Keywords: bronchoscopy; endoscopy; patient reported outcome measures
MeSH Terms: conditions — Bronchial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Bronchoscopy under local anesthesia: Bronchoscopy under local anesthesia
  Interventions: Other: no intervention
- Bronchoscopy under anxiolysis: Bronchoscopy under anxiolysis
  Interventions: Other: no intervention
- Bronchoscopy under conscious sedation: Bronchoscopy under conscious sedation
  Interventions: Other: no intervention
- Bronchoscopy under general anesthesia: Bronchoscopy under general anesthesia
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — only observational

SUMMARY:
'Patient-reported outcomes' (PROMS) and 'patient-reported experiences' (PREMS) are increasingly important parameters in evaluating and adjusting clinical procedures and strategies in healthcare.

Validated disease-specific PROMS related to bronchoscopic procedures are not available and examples in the medical literature are very scarce.

DETAILED DESCRIPTION:
The potential usefulness of PROM/PREMS is multiple:

1. Quality improvement within the current clinical care structure
2. Monitoring the health status of the population
3. Contribution to decision-making regarding financing of care
4. Increase employee and patient involvement in clinical care pathways
5. Rationalize the deployment of medical personnel and resources
6. Integration of data in electronic patient files and registers

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Patient referred for diagnostic flexible bronchoscopy
* Procedure performed in outpatient setting

Exclusion Criteria:

* Patient unable to adequately respond to the contents of the patient questionnaire.
* Procedure performed in hospitalised setting
* Patient with active pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Out-of-hospital care
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Procedure-related dyspnea scale (VAS) | 24 hours
  Procedure-related dyspnea scale (VAS)
Procedure-related pain scale (VAS) | 24 hours
  Procedure-related pain scale (VAS)
Procedure related cough scale (VAS) | 24 hours
  Procedure related cough scale (VAS)
General patient satisfaction | 24 hours
  General patient satisfaction VAS scale

SECONDARY OUTCOMES:
Procedure-related complications: | 24 hours
  bleeding + grading; pneumothorax; hypoxaemia; hypercapnia; respiratory rate; heart rate.
Sedation-related complications | 24 hours
  paradoxical agitation; GCS; hypoxaemia; hypercapnia
Diagnostic yield | 30 days
  number of biopsies; histological diagnosis; DNA extraction.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Yserbyt, MD, PhD, Principal Investigator — MD
Locations (1):
- VITAZ, Sint-Niklaas, Belgium

IPD SHARING:
Plan to Share IPD: No